CLINICAL TRIAL: NCT05291923
Title: Predictors of Severity of Postoperative Pancreatic Fistula After Pancreatoduodenectomy.
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-POPF-01
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pancreatic Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post whipple's procedure patients
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Pancreaticoduodenectomy is one of the commonly performed procedure for periampullary carcinoma/distal cholangio carcinoma/head of pancreas carcinoma. Postoperative pancreatic fistula remains the most important postoperative complication following pancreatic surgery. It's severity ranges from biochemical leak to grade C POPF which can lead to mortality. Radiological and biochemical parameters in early postoperative period predicts the severity of POPF after pancreatoduodenectomy. In this study, we will be evaluating the biochemical parameters and imaging findings as predictors of the severity of postoperative pancreatic fistula after pancreatoduodenectomy in early postoperative period.

DETAILED DESCRIPTION:
(a) Aim and Objective - The aim of this study is to evaluate the biochemical parameters and imaging findings as predictors of the severity of postoperative pancreatic fistula after pancreatoduodenectomy in early postoperative period

Methodology:

1. Study population: All those operated for pancreatoduodenectomy during the period of December 2021 to May 2023 will be enrolled in this study, meeting the inclusion and exclusion criteria. On an average 3-4 cases are operated per month in ILBS.
2. Study design: Prospective observational study.
3. Study period: From the date of clearance by the Institutional Ethics Committee, till May 2023.
4. Sample size with justification: All consecutive patients undergoing pancreatoduodenectomy for the above-mentioned study period (expected sample size 40)
5. Intervention: none.
6. Monitoring and assessment:

1) Definitions: International study group on pancreatic fistula definition of Post-Operative Pancreatic Fistula POPF) will be used which are as follows: drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content greater than 3 times the serum amylase activity

Variables to be assessed:

Patient characteristics - Age, Sex, Height, Weight, BMI, Serum albumin levels, Pancreatic parenchymal thickness- at spleno-portal confluence, Indication of Pancreatoduodenectomy -Peri ampullary mass, head of pancreatic mass, distal cholangiocarcinoma Operative Parameters - Duration of surgery, Blood Loss, Pancreatic consistency, Intraoperative remnant pancreatic parenchymal thickness at pancreatojejunostomy site/ spleno portal confluence.

Postoperative measurements -

1. Drain Fluid amylase (POD 1,3 & 5) & serum amylase
2. Serum Procalcitonin, C-reactive protein and albumin (POD 5)
3. Remnant pancreatic parenchymal thickness & change in thickness at pancreaticojejunostomy site/splenoportal confluence on NCCT abdomen (POD 5)
4. Presence & location of intra-abdominal collection by NCCT abdomen (POD 5)
5. Interventions required if any for management of complications

Statistical Analysis: Data will be entered into Excel Worksheet and statistical analyses will be performed by SPSS Statistics version 22 (IBM Corp., Armonk, NY). Statistical data will be represented as frequencies (%) where the continuous variables will be expressed as medians and interquartile range (IQR). Continuous variables will be compared with the student t test and Mann-Whitney test as appropriate. Differences between proportions derived from categorical data will be compared with Chi-square or Fischer's exact test. Variables will be correlated with clinical outcomes. ROC curve will be used for biochemical markers and imaging findings Repeated analyses of measures will be applied wherever applicable.

Adverse effects: None

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing Pancreatoduodenectomy at ILBS
* Duct to mucosa pancreaticojejunostomy

Exclusion Criteria:

* Refused for consent
* Age < 18 yrs
* Hepatopancreatoduodenectomy
* Multi-visceral resection
* Re-exploration before POD 5
* Pancreaticogastrostomy
* Dunking type of pancreaticojejunostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing pancreatoduodenectomy at ILBS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
change in pancreatic parenchymal thickness at pancreaticojejunostomy site/spleno-portal confluence on postoperative day 5 predicts the severity of postoperative pancreatic fistula after pancreatoduodenectomy in early postoperative period | Post operative day 5

SECONDARY OUTCOMES:
Levels of C-reactive protein among the different grades of post operative pancreatic fistula | Post operative day 5
Levels of serum albumin among the different grades of postoperative pancreatic fistula. | Post operative day 5
Levels of serum procalcitonin among the different grades of postoperative pancreatic fistula. | Post operative day 5
Intra-abdominal collection among the different grades of postoperative pancreatic fistula by NCCT abdomen. | Post operative day 5
Location of intra-abdominal collection among the different grades of postoperative pancreatic fistula by NCCT abdomen. | Post operative day 5

CONTACTS AND LOCATIONS:
Overall Officials: Dr Piyush Kumar Sinha, MCh, Study Director — Institute of Liver and Biliary Sciences, New Delhi
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No